CLINICAL TRIAL: NCT00138060
Title: Protocole Evaluant Chez Des Patients Porteurs de Cancers Colorectaux Metastatiques l'Interet Des Determinants Genotypiques Pour l'Optimisation de l'Efficacite et de la Tolerance de la Chimiotherapie Par Irinotecan et 5-fluorouracile
Brief Title: Toxicity/Benefit Ratio Optimization of Chemotherapy in Colorectal Cancer (CRC) Patients by Determination of Individual Genotypic Determinants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche Clinique sur les Cancers et le Sang (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Gilles Freyer, IRCCSang
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLOGEN
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: genotypic profile; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: irinotecan — 180 mg/m² or 260 mg/m² in 90 minutes every 15 days
Drug: 5 fluorouracil — 400 mg/m² in bolus in day 1 and 2400 mg/m² in 46 hours perfusion

SUMMARY:
This study intends to optimize a fluorouracil/irinotecan chemotherapy regimen by the identification of individual thymidylate synthase (TS) and UDP-glucuronosyltransferase 1 (UGT1A1) polymorphisms before the first administration.

The results of this identification determine the chemotherapy type: high-dose irinotecan or not.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time without prejudice
* Ages between 18 and 85 years
* Histologically confirmed colorectal cancer
* No treatment for metastatic disease
* No irinotecan previously administered
* World Health Organization (WHO) performance status < 3
* Laboratory values :

  * neutrophils > 1.5 x 10^9/L;
  * platelet count > 100 x 10^9/L;
  * serum creatinine < 130µmol/L;
  * serum bilirubin < 2 x upper limit of normal (ULN);
  * ASAT and ALAT < 2.5 x ULN;
  * alkaline phosphatase < 5 x ULN.
* At least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) criteria

Exclusion Criteria:

* History of another malignancy except cured basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix, breast or bladder.
* Other concomitant anticancer therapy.
* Pregnant or lactating women.
* Women of childbearing potential unless using a reliable and appropriate contraceptive method.
* Symptomatic cerebral or leptospiral metastasis.
* Intestinal obstruction.
* Uncontrolled seizures (diabetes, severe infection).
* Clinically significant cardiac disease.
* Central nervous system disorders or severe psychiatric disability.
* Participation in any investigational study within 4 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
tumor response rate | during the treatment

SECONDARY OUTCOMES:
toxicity | during the treatment
pharmacokinetics | during the first administration

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Freyer, MD, Principal Investigator — Department of Oncology, CHLS, 69310 Pierre Benite, France
Locations (6):
- France (6):
  - Department of Oncology, CHU, Grenoble
  - Department of Oncology, IPC, Grenoble
  - Department of Gastroenterology, CHLS, Pierre-Bénite
  - Department of Oncology - CHLS, Pierre-Bénite
  - Department of Oncology, ICL, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- [Background] Iyer L, Das S, Janisch L, Wen M, Ramirez J, Karrison T, Fleming GF, Vokes EE, Schilsky RL, Ratain MJ. UGT1A1*28 polymorphism as a determinant of irinotecan disposition and toxicity. Pharmacogenomics J. 2002;2(1):43-7. doi: 10.1038/sj.tpj.6500072. PMID 11990381